CLINICAL TRIAL: NCT03264963
Title: Upper Airway Training for Treatment of Snoring Using Smartphone Application
Brief Title: Upper Airway Training for Treatment of Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: UMN Medical Devices Center (Unknown); Fairview Sleep Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1606S88671
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Snoring
Keywords: Upper airway exercises; Smart phone application
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Control
- Intervention (Experimental)
  Interventions: Other: Smart phone game play

INTERVENTIONS:
Other: Smart phone game play — Voice controlled smart phone game play 15 minutes daily and recording sounds of sleep environment 2 night per week for 12 weeks
  Arms: Intervention
Other: Control — Recording of sleep environment 2 nights per week for 12 weeks
  Arms: Control

SUMMARY:
The objective of this study is to reduce the incidence or intensity of snoring in a patient population of known simple snorers without sleep apnea using smartphone based application which allows participants to play voice controlled games using various articulations resulting in tongue base movements.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent in English.
2. Age is between 20 and 65.
3. BMI less than 32
4. Less than 5% variance in weight since sleep study.
5. Snoring without health risk related to sleep apnea and not currently receiving treatment.

   1. Mild OSA or negative HSAT or PSG within past year with AHI 0-14
   2. Has refused oral appliances, CPAP, weight loss, surgery or positional therapy.
6. Owns an iPhone 4 or newer and is comfortable downloading and using apps.
7. Complaint of habitual snoring 3 or more nights per week
8. Rated by polysomnograph technologist as moderate or loud snoring.

Exclusion Criteria:

1. Non-fluent in English.
2. Persistent rhinitis diagnosis or nasal obstruction.
3. BMI > 32
4. Greater than 5% variance in weight since sleep study.
5. Diagnosis of moderate to severe sleep apnea or any other sleep disorder (insomnia, RLS)
6. Insufficient sleep, defined as getting fewer than 6 hours of sleep on an average night based on self report.
7. Spouse/partner is also a habitual snorer.
8. Lacking ability to consent for themselves.
9. Heavy drinker (self reported average more than 2 drinks per day).
10. Regular narcotics (greater than 3 times/week)
11. Epworth sleepiness scale score > 11 or one near miss accident in the past 6 months.
12. Medical conditions as follows: symptomatic cardiopulmonary disease, chronic renal insufficiency, poorly controlled mental illness.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-05-18 (Actual)

PRIMARY OUTCOMES:
Snoring Intensity | 12 weeks
  Snoring sounds >60 db
Snoring Rate | 12 weeks
  Snoring sounds/hour of sleep

SECONDARY OUTCOMES:
Sleep Quality | 12 weeks
  Self reported sleep quality on likert scale (0 to 5)
Bed Partner Sleep Quality | 12 weeks
  Bed partner reported sleep quality on likert scale (0 to 5)
Sleepiness | 12 weeks
  Epworth sleepiness score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goswami U, Black A, Krohn B, Meyers W, Iber C. Smartphone-based delivery of oropharyngeal exercises for treatment of snoring: a randomized controlled trial. Sleep Breath. 2019 Mar;23(1):243-250. doi: 10.1007/s11325-018-1690-y. Epub 2018 Jul 21. PMID 30032464